CLINICAL TRIAL: NCT01743963
Title: Intervention to Increase Screening for Glucocorticoid Induced Diabetes
Acronym: CDA-GID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Liron Caplan MD, PhD, Associate Professor, VA Eastern Colorado Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 176843
Record Dates: First submitted 2012-11-20; First posted 2012-12-06 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus
Keywords: efficacy; glucocorticoid
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Support Intervention (Experimental): Clinical pharmacists mediated computerized decision support
  Interventions: Behavioral: Decision support
- Usual Care (Active Comparator): Clinicians' typical approach for GID monitoring
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Decision support — Clinical pharmacists mediated computerized decision support
  Arms: Decision Support Intervention
Behavioral: Usual Care — clinicians typical apporach for GID monitering
  Arms: Usual Care

SUMMARY:
Using glucocorticoid induced diabetes (GID) we will conduct a small feasibility randomized intervention trial to improve GID management for veterans who are prescribed chronic glucocorticoids. Approximately 20 primary care providers (caring for approximately 100 veterans on chronic steroids) will receive decisional support (automatically-derived orders for hemoglobin A1C, to be co-signed by providers). Approximately 20 providers (caring for 100 veterans) who did not receive decisional support will serve as the control population. We will measure the time from randomization until the provider signs an order for hemoglobin A1C for both groups. The trial will be conducted at the VA's Eastern Colorado Health Care System (ECHCS) and will last approximately 6 months. After the completion of the trial for each provider, we will conduct a brief interview and survey of the participating providers to assess the acceptability of decisional support interventions to manage GID [protocol, page 1-2]. No patient data (PHI) will be collected by the providers.

DETAILED DESCRIPTION:
Aim 1: Conduct a single site randomized controlled feasibility trial of a decisional support intervention to reduce ADRLLS by improving providers' adherence to GID prevention measures. Approximately 20 primary care providers (caring for approximately 100 veterans on chronic steroids who have not been screened for diabetes in the last year) will be randomly assigned to receive decisional support for GID prevention measures (automatically-derived orders for hemoglobin A1C, to be co-signed by providers). These providers will be compared with 20 providers (caring for 100 veterans not screened for diabetes in the last year) who are randomly assigned to not receive decisional support for management of GID (i.e. the control group). The trial will be conducted at the VA's Eastern Colorado Health Care System (ECHCS) and will last approximately 6 months. Study administration will be coordinated through the Colorado Research Award Enhancement Program (Colorado REAP).

Aim 1a) Procedural Endpoints: As a feasibility trial, this study includes multiple procedural endpoints, such as provider participation rates, to assess the viability of the intervention, rather than a single primary efficacy outcome measure (for details, pages 6-7).

Aim 1b) Preliminary Estimates of Efficacy: We will determine the Delay Interval-the number of days from when a provider is randomized until the provider orders the GID prevention measure. Use of this continuous measure will maximize the power of this feasibility study, though we will also determine proportions of patients for whom these measures were ordered at six months, so that we may estimate the sample size for a subsequent multi-center randomized control trial.

Aim 1c) Post-trial de-briefing: Using structured interviews, we will examine the opinions of providers after they have participated in the GID feasibility trial, in order to gather additional qualitative data regarding the ADRLL framework and refine the intervention for a subsequent randomized controlled trial. Providers will also complete a brief survey assessing their preference for the intervention.

ELIGIBILITY:
Inclusion criteria:

* Must be 18-90 years old
* Must be served by the ECHCS VA sytem
* Must have chronic glucocorticoid exposure (greater than or equal to 90 days of oral glucocorticoids)
* Eligible providers will consist of those primary care practitioners within the ECHCS with at least one patient meeting the above criteria. For each veteran, the primary care provider (PCP) will be defined as the patient's current general internal medicine or family practice practitioner. In the rare instance in which the patient has no PCP within the VA system, the specialist with the greatest number of patient encounters during the past 12 months will be eligible for inclusion. For every patient, only one provider will be randomized (to avoid multiple exposure to the intervention for some patients). The consent procedure is described below.

Exclusion Criteria:

* Veterans who have had a hgbA1C test within the previous 12 months will be excluded.
* Providers without eligible patients (described above), will be excluded.
* Providers declining to give consent will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liron Caplan, MD, PhD, Principal Investigator — Veteran Affairs
Locations (1):
- Liron Caplan, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decision Support Intervention | Usual Care
Started | 21 | 17
Completed | 21 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Support Intervention | Usual Care | Total
Number analyzed (Participants) | 21 | 17 | 38
Age, Customized [Number; unit: participants] — We were not authorized by the IRB to record this information; however, all participants were between the ages of 18 and 90, as specified in the inclusion criteria.
  participants
    18 to 90 years | 21 | 17 | 38
Sex: Female, Male [Count of Participants; unit: Participants] — We were not authorized by IRB to record this information.
  Participants
    Female | NA — We were not authorized by IRB to record this information. | NA — We were not authorized by IRB to record this information. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — We were not authorized by IRB to record this information. | NA — We were not authorized by IRB to record this information. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Delay Interval (Days From Randomization Until the Provider Signs the Order for a hgbA1C Level).
Description: For follow-up laboratory data within the VA system, adherence will be monitored through prospective accrual of administrative data and review of the medical record. Results will be reported as the proportion receiving the preventive measure versus time, i.e. with Kaplan-Meier plots. We will then determine the variance of Delay Interval. For the preliminary measure of efficacy, the Delay Interval will be compared between patients whose providers were assigned to the intervention and patients whose providers did not receive the intervention.
Time Frame: 6 MONTHS
Population: 21 patients cared for by 6 providers in intervention arm; 17 patients cared for by 6 providers in usual care arm.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Decision Support Intervention | Usual Care
Number analyzed (Participants) | 21 | 17
Days | 12 [6.3 to 398.7] | 104 [6.3 to 398.7]

2. Secondary Outcome: Feasibility/Reach/Adoption
Description: Measurements of intervention delivery include recruitment numbers and provider Participation Rates for enrollment and retention. The definition of study feasibility consists of provider enrollment rates >= 50%. Results reported using descriptive statistics (proportions, means, standard deviations, and ranges).
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Feasibility/Reach/Adoption
Description: Measurements of intervention delivery include the "representativeness" of providers (differences between participants/non-participants). Results reported using descriptive statistics (proportions, means, standard deviations, and ranges).
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Feasibility/Reach/Adoption
Description: Measurements of intervention delivery include the rationale used by clinicians declining participation. Results reported using descriptive statistics (proportions, means, standard deviations, and ranges).
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Feasibility/Reach/Adoption
Description: Measurements of intervention delivery include numbers of veterans excluded from the intervention. Results reported using descriptive statistics (proportions, means, standard deviations, and ranges).
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Entire duration of study
Description: No adverse events were observed.
Arm/Group | Decision Support Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/17
Other Adverse Events (participants affected / at risk) | 0/21 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No